CLINICAL TRIAL: NCT01684189
Title: A Non-interventional Prospective Registry to Monitor the Events of Febrile Neutropenia and Invasive Fungal Infections and the Diagnostic and Therapeutic Management in Patients With Malignant Hematologic Diseases After Chemotherapy
Brief Title: Registry of Febrile Neutropenia and Invasive Fungal Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MISP38887
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2011-11

CONDITIONS: Hematological Disease; Febrile Neutropenia; Fungal Infections
MeSH Terms: conditions — Hematologic Diseases; Febrile Neutropenia; Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient registry: Patients with newly diagnosed malignant hematological diseases will be enrolled into this registry
  Interventions: Other: Patient registry

INTERVENTIONS:
Other: Patient registry — Patient registry without study intervention

SUMMARY:
Objectives：

1. To assess the percentage of febrile neutropenia and suspected fungal-related febrile episodes in patients receiving chemotherapy
2. To explore the percentage/distribution of infectious origins of febrile neutropenia
3. To explore the percentage/distribution of infectious pathogens of febrile neutropenia
4. To explore clinical outcomes of different infectious origins/pathogens in febrile neutropenia episodes
5. To have a clear view of therapeutic actions in the management of hematological patients with febrile neutropenia and suspected fungal-related febrile episodes

DETAILED DESCRIPTION:
Objectives：

1. To assess the percentage of febrile neutropenia and suspected fungal-related febrile episodes in patients receiving chemotherapy
2. To explore the percentage/distribution of infectious origins of febrile neutropenia
3. To explore the percentage/distribution of infectious pathogens of febrile neutropenia
4. To explore clinical outcomes of different infectious origins/pathogens in febrile neutropenia episodes
5. To have a clear view of therapeutic actions in the management of hematological patients with febrile neutropenia and suspected fungal-related febrile episodes

Study Design：

* This is a single institute, prospective, non-interventional registry for monitoring events of febrile neutropenia in hematological patients
* Patients with newly diagnosed malignant hematological diseases will be enrolled into this registry

Study Procedures： Data collection will include patients' basic information, underlying disease, baseline blood chemistry and blood cell counts, antifungal prophylaxis, C/T regimens, neutrophils and other blood cells, fever diagnosis and infectious sites work-up, clinical response, microbiology (including bacteria and fungus culture), renal and liver function, clinical diagnosis, work-up and intensive procedures and results, antifungal and antibacterial agents (including dosage, duration, and route), other drugs used (including antivirals, antineoplastics, corticosteroids, immunomodulators), clinical significant changes

Sample Size Calculation and Statistical Analysis： Approximately 100 febrile neutropenia episodes in 500 chemotherapy cycles will be collected. This is an observational and exploratory study without hypothesis tests. Study subjects will be collected and monitored under normal clinical practice, and the sample size will be limited due to the hospital scale and disease characteristic (the sample size calculation is inapplicable here). All evaluations will be shown by exploratory and descriptive data analysis. The number of cases for each investigative definition, the corresponding percentage and the 95% confidence interval will be described.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new diagnosed hematological diseases (acute and chronic myeloid and lymphoid leukemia, multiple myeloma, non-Hodgkin's and Hodgkin's lymphoma, myelodysplastic syndromes)
* Patients who are receiving chemotherapy and have ongoing febrile episodes

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed malignant hematological diseases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chung Wang, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan